CLINICAL TRIAL: NCT03107949
Title: Percutaneous Temporary Placement of a Phrenic Nerve Stimulator for Diaphragm Pacing
Brief Title: Percutaneous Temporary Placement of a Phrenic Nerve Stimulator for Diaphragm Pacing (RESCUE1)
Acronym: RESCUE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lungpacer Medical Inc. (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P-100; G170057 (Other: FDA)
Record Dates: First submitted 2017-03-21; First posted 2017-04-11 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Ventilator Induced Diaphragm Dysfunction
Keywords: Diaphragm atrophy; VIDD; weaning failure; SBT

STUDY DESIGN:
Intervention Model Description: LIVE Catheter is temporarily insertied into the left subclavian vein and connected to the LCU for DPTS to be delivered daily. The DPTS includes the LIVE Catheter, LCU and intermediate cable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lungpacer Diaphragm Pacing Therapy (DPTS) (Experimental): The LIVE Catheter will be temporarily inserted (LIVE Catheter will be inserted into every patient enrolled and can stay in place for up to 30 days) into the left subclavian vein and connected to the Lungpacer Control Unit in order to perform diaphragm pacing to stimulate the phrenic nerves and activate the diaphragm 3 x a day on all patients until extubated/removed from mechanical ventilation or until day 30 whichever comes first.
  Interventions: Device: Lungpacer DPTS (Diaphragm Pacing Therapy System)

INTERVENTIONS:
Device: Lungpacer DPTS (Diaphragm Pacing Therapy System) — Lungpacer Diaphragm Pacing therapy (DPTS) will be conducted in daily sessions until the patient has been extubated or day 30 if not extubated.
  Other Names: LIVE Catheter; RESCUE 1

SUMMARY:
An early feasibility study to investigate the safety and feasibility of the Lungpacer Diaphragm Pacing Therapy System (DPTS) as a therapy to recondition and strengthen the diaphragm of patients who have been intubated and invasively mechanically ventilated for > or = 7 days, have failed two or more spontaneous breathing trials (SBT), and were not hypervolemic during the latest SBT.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a life saving technology but can also cause damage to the lungs and diaphragm such as ventilator induced diaphragmatic dysfunction (VIDD). Research has shown that after being on mandatory MV and sedated the diaphragm begins to atrophy within as little as 18 hours. The DPTS is a temporary therapy that consists of the Lungpacer IntraVenous Electrode Catheter (LIVE Catheter) and the lungpacer Control Unit (LCU) system. The LIVE Catheter is a proprietary central venous catheter that incorporates pacing electrodes in strategic areas that align with the left and right phrenic nerves in order to stimulate the nerves to recruit the diaphragm. The LIVE Catheter can also be used for fluid delivery like any other central venous catheter. This early feasibility trial will investigate the safety and feasibility of the DPTS as a therapy to recondition and strengthen the diaphragm by stimulating the diaphragm through daily sessions so the patient may be more quickly liberated from MV. The patient population includes those who have been mechanically ventilated for > or = to 7 days, have failed two or more SBTs, and were not hypervolemic during the latest SBT. Patients must have resolution of the initial indication for placement on MV before entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* have been mechanically ventilated for > or = 7 days and have not met criteria for successful weaning during this period; and
* have failed at least two SBTs, one of which is the study specific SBT. (Self-extubation with subsequent reintubation within 48 hours is considered a failed SBT).

Exclusion Criteria:

* currently on extracorporeal membrane oxygenation (ECMO);
* weaning failure due to hypervolemia;
* known anatomy that prevents insertion of the LIVE Catheter into the left subclavian vein;
* history of congenital heart disease;
* clinically overt congestive heart failure;
* pre-existing neuromuscular diseases that could affect the respiratory muscles;
* pleural effusions occupying greater than one third of the pleural space on either side;
* BMI > or = 40;
* known or suspected phrenic nerve paralysis;
* any electrical device (implanted or external) that may be prone to interaction with or interference from the Lungpacer DPTS including neurological pacing/stimulator devices, cardiac pacemakers and defibrillators;
* bacteremia (blood cultures must be negative for 48 hours);
* current haemodynamic instability, shock or severe sepsis;
* terminally ill with 6 months or less life expectancy or not committed to full care;
* known or suspected to be pregnant or lactating; and
* actively participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Successful Placement of the LIVE Catheter | You will undergo an evaluation immediately following the LIVE Catheter insertion procedure to confirm that the LIVE Catheter has been successfully placed in the correct position in your vein.
  Successful placement of the LIVE Catheter via the Left Subclavian vein at the initiation of study will be assessed by placement confirmation via Chest Xray
Capture of phrenic nerve | Measured during daily Diaphragm Pacing Therapy sessions from time of LIVE Catheter insertion to time of extubation or day 30 whichever comes first
  Successful capture and stimulation of at least one phrenic nerve as assessed by the change in the ventilator waveform and or diaphragm contraction.
Diaphragm contraction noted upon stimulation of the phrenic nerve | Measured during daily Diaphragm Pacing Therapy sessions from time of LIVE Catheter insertion to time of extubation or day 30 whichever comes first.
  Demonstration of the ability to contract the diaphragm via phrenic nerve stimulation will be evaluated by palpation of the diaphragm or visualization of the ventilator waveform change.
Removal of LIVE Catheter | Removal of LIVE Catheter will occur 2 days after extubation or on day 30 if subject has not been extubated.
  Successful removal of the LIVE Catheter two days after date of extubation but before the end of the study on day 32

OTHER OUTCOMES:
Evaluation of SAE's related to the use of the LIVE Catheter | From enrollment and insertion of the LIVE Catheter through LIVE Catheter removal or day 30 whichever comes first.
  All SAE's related to the use of the LIVE Catheter will be evaluated to assess a reasonable safety profile associated with the LIVE Catheter insertion and removal procedure and the use of the DPTS in all study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Clark, RN, BSN, Study Director — Vice Presdient of Clinical Affairs, Lungpacer Medical, Inc.
Locations (4):
- United States (4):
  - University of Florida Health Science Center - Shands, Gainesville, Florida
  - New York University Medical Center, New York, New York
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Only investigators participating in this clinical trial will be able to see final de-identified participant data at the completion of the study and it will be available through Syntactx.